CLINICAL TRIAL: NCT02018848
Title: Internet-delivered Attention Training for Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humboldt-Universität zu Berlin (Other)
Responsible Party: Principal Investigator, Dr. Andrea Ertle, Dr. phil. Dipl. Psych., Humboldt-Universität zu Berlin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HU-ATP-OCD-2013
Record Dates: First submitted 2013-11-28; First posted 2013-12-23 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Attention Training; Attention Bias Modification; Dot-Probe Task; Randomized Controlled Trial; Online Treatment; Washing; Checking
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Adenosine Triphosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Attention Training Placebo (Placebo Comparator): Same procedure, stimulus material, frequency and duration as in experimental group.
  The only difference: In the placebo group the probe randomly appears at one of the two locations on the screen so as not to train attention in any direction.
  Thus, the placebo training sessions are identical to the bias assessment sessions.
- Attention Training Program (Experimental): The Attention Training consists of a modified dot-probe task. In this task pairs of pictures (OCD-relevant/neutral) are presented for 500 ms on a computer screen. Next, a probe appears on one of the two former picture locations. Participants have to react to that probe by pressing the corresponding button on the keyboard. One training session takes approximately 10 minutes in which 160 stimulus pairs are shown.
  In the experimental group the probe always appears at the location of the neutral picture so as to train attention away from OCD-relevant stimuli.
  Participants are asked to complete at least 2 training sessions per week over a period of 5 weeks. The first and last session are bias assessment sessions (see outcome measures), but participants stay blind to this.
  Interventions: Behavioral: Attention Training Program

INTERVENTIONS:
Behavioral: Attention Training Program
  Other Names: ATP; Attention Bias Modification Treatment; ABMT; Bias Modification; Attentional Training
  Arms: Attention Training Program

SUMMARY:
The goal of this study is to investigate an attention training program for participants with Obsessive-Compulsive Disorder. The attention training consists of a modified dot probe task with picture stimuli related to washing and checking paired with neutral pictures.

Participants are randomly assigned to an experimental and a placebo-control group. After a minimum of 4 weeks of attention training we expect to find differences between participants of the experimental and the control group in terms of attention bias, OCD symptoms, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary OCD according to OCI-R self report (cut-off >=18)

Exclusion Criteria:

* suicidal
* substance abuse or addiction
* psychotic symptoms
* visual impairment if not compensated with optical aid

Current treatment is not an exclusion criterion, but data on treatment status (current psycho- or pharmacotherapy for OCD) will enter our statistical analyses.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale Self-Report Scale (Y-BOCS-SRS) T1 | pre-treatment, estimated: between day 1 and day 7 after enrolment (no time limit set)
  The Y-BOCS-SRS measures severity of OCD symptoms.
Yale-Brown Obsessive-Compulsive Scale Self-Report Scale (Y-BOCS-SRS) T2 | post-treatment, between day 1 and 6 after T2 Bias Assessment (time limit set)
  The Y-BOCS-SRS measures severity of OCD symptoms.
Yale-Brown Obsessive-Compulsive Scale Self-Report Scale (Y-BOCS-SRS) T3 | follow-up, between day 27 and 50 after T2 questionnaires (time limit set)
  The Y-BOCS-SRS measures severity of OCD symptoms.

SECONDARY OUTCOMES:
Obsessive-Compulsive Inventory-Revised (OCI-R) T1 | pre-treatment, estimated: between day 1 and day 7 after enrolment (no time limit set)
  The OCI-R measures severity of OCD symptoms.
Obsessive-Compulsive Inventory-Revised (OCI-R) T2 | post-treatment, between day 1 and 6 after T2 Bias Assessment (time limit set)
  The OCI-R measures severity of OCD symptoms.
Obsessive-Compulsive Inventory-Revised (OCI-R) T3 | follow-up, between day 27 and 50 after T2 questionnaires (time limit set)
  The OCI-R measures severity of OCD symptoms.

OTHER OUTCOMES:
Beck Anxiety Inventory (BAI) T1 | pre-treatment, estimated: between day 1 and day 7 after enrolment (no time limit set, all further steps relative to exact time point of T1 questionnaires)
  The BAI measures severity of anxiety symptoms.
Beck Anxiety Inventory (BAI) T2 | post-treatment, between day 1 and 6 after T2 Bias Assessment (time limit set)
  The BAI measures severity of anxiety symptoms.
Beck Anxiety Inventory (BAI) T3 | follow-up, between day 27 and 50 after T2 questionnaires (time limit set)
  The BAI measures severity of anxiety symptoms.
Beck Depression Inventory II (BDI-II) T1 | pre-treatment, estimated: between day 1 and day 7 after enrolment (no time limit set, all further steps relative to exact time point of T1 questionnaires)
  The BDI measures severity of depressive symptoms.
Beck Depression Inventory II (BDI-II) T2 | post-treatment, between day 1 and 6 after T2 Bias Assessment (time limit set)
  The BDI measures severity of depressive symptoms.
Beck Depression Inventory II (BDI-II) T3 | follow-up, between day 27 and 50 after T2 questionnaires (time limit set)
  The BDI measures severity of depressive symptoms.
Attention bias towards OCD-relevant stimuli at T1 measured with a dot-probe task. | after T1 questionnaires and pre-treatment, estimated: between day 1 and 3 after T1 questionnaires (no time limit set)
  Attention bias is measured using a dot-probe task. In this task pairs of pictures (OCD-relevant/neutral) are presented briefly on a computer screen. Next, a probe randomly appears on one of the two former picture locations. Participants have to react to that probe by pressing the corresponding button on the keyboard.
  Attention bias is calculated as the mean difference in reaction times between trials in which the probe appears at the OCD-relevant location vs. trials in which it appears at the neutral location. The bias assessment session is masked as first training sessions in both groups.
Attention bias towards OCD-relevant stimuli at T2 measured with a dot-probe task. | post-treatment, after a minimum of 8 training sessions over a time of 4 weeks, estimated: between day 1 and 4 after last training session (no time limit set)
  Attention bias is measured using a dot-probe task. In this task pairs of pictures (OCD-relevant/neutral) are presented briefly on a computer screen. Next, a probe randomly appears on one of the two former picture locations. Participants have to react to that probe by pressing the corresponding button on the keyboard.
  Attention bias is calculated as the mean difference in reaction times between trials in which the probe appears at the OCD-relevant location vs. trials in which it appears at the neutral location.

CONTACTS AND LOCATIONS:
Locations (1):
- Humboldt-Universität zu Berlin, Berlin, State of Berlin, Germany